CLINICAL TRIAL: NCT06563258
Title: Efficacy of Biodex Balance Training Versus Whole Body Vibration Training in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, walaa, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005293
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A Prospective parallel group single-blind randomized control trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Whole Body Vibration Training in Patients With Knee Osteoarthritis (Experimental): Group A Will receive WBV Training with frequency of 35 Hz, peak-to-peak amplitude of 4- to 6-mm Vertical sinusoidal vibration, and the total exposure time of 30 minutes (vibration 60 seconds, interval rest 60 seconds) in addition to traditional exercises,3 sessions per week for four weeks.
  Interventions: Device: A vibration device; Other: traditional exercises
- Biodex Balance Training in Patients With Knee Osteoarthritis (Experimental): Group B will receive Biobex training, Total time of training was 10 minutes each set is 3 minutes with 20-second rest intervals in addition to traditional exercises,3 sessions per week for four weeks.
  -
  Interventions: Device: Biodex Balance Training
- traditional exercises in Patients With Knee Osteoarthritis (Experimental): Group C Patients will receive only traditional exercises, 3 sessions per week for four weeks. a good general guideline is 2-3 sets of 10-15 repetitions for each exercise.
  Interventions: Other: traditional exercises

INTERVENTIONS:
Device: Biodex Balance Training — Sixty Subjects of both genders aged 40-60 years old with grade 2 knee osteoarthritis years will diagnosed by orthopedists they will assigned randomly into three groups:
  * Group A Will receive WBV Training with frequency of 35 Hz, peak-to-peak amplitude of 4- to 6-mm Vertical sinusoidal vibration, and the total exposure time of 30 minutes (vibration 60 seconds, interval rest 60 seconds) in addition to traditional exercises,3 sessions per week for four weeks. , A vibration device (My7™ model Personal Plate, Power Plate, Northbrook, IL, USA) will used in all WBVT sessions.
  * Group B will receive Biobex training and traditional exercises Total time of training was 10 minutes each set is 3 minutes with 20-second rest intervals
  * Group C Patients will receive only traditional exercises, 3 sessions per week for four weeks. a good general guideline is 2-3 sets of 10-15 repetitions for each exercise.
  Arms: Biodex Balance Training in Patients With Knee Osteoarthritis
Device: A vibration device — WBV Training with frequency of 35 Hz, peak-to-peak amplitude of 4- to 6-mm Vertical sinusoidal vibration, and the total exposure time of 30 minutes (vibration 60 seconds, interval rest 60 seconds) in addition to traditional exercises,3 sessions per week for four weeks. , A vibration device (My7™ model Personal Plate, Power Plate, Northbrook, IL, USA) will used in all WBVT sessions.
  Arms: Whole Body Vibration Training in Patients With Knee Osteoarthritis
Other: traditional exercises — 1. Stretch exercises (flexibility exercise) Rectus femoris, Iliotibial band, Hamstring and self-stretch for calf muscle (3sets, each stretch 30 sec hold, between each set 5sec rests).
  2. Strengthen exercises(resistance exercise)
     1. Isometric Exercises for quadriceps (10 rep,3sets)
     2. Hip abductors strengthening 45 degree (10 rep,3sets)
     3. Hip extensor strengthening 15 degree (10 rep,3sets)
     4. Straight leg raising 45-70 degree (10 rep,3sets)
     5. Short arc knee extension (10 rep,3sets)
  Arms: Whole Body Vibration Training in Patients With Knee Osteoarthritis; traditional exercises in Patients With Knee Osteoarthritis

SUMMARY:
This study will be conducted to answer the research question:

Are there differences between the effect of Biodex balance training and Whole-body vibration training on Knee osteoarthritis?

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of biodex training balance versus whole body vibration training on Knee osteoarthritis on:

* Pain intensity
* static balance
* dynamic balance
* Functional ability level

ELIGIBILITY:
Inclusion criteria:

1. Subjects age between (40-60) years old.
2. Radiologic findings had to be compatible with knee OA grade 2 in a simple X ray.
3. Tenderness on medial tibial plateau
4. Intensity of pain: visual analogue scale equal to 5 or greater
5. Failure of two or more types of previous conservative treatment (medication, anti-inflammatory drugs, physical therapy, stretching, acupuncture, orthotics and others) in the last three months

Exclusion Criteria:

1. Neurological and vestibular system disorder, systematic inflammatory disease, steroid injections in the last six months
2. Subjects with diabetes mellitus.
3. acute symptomatic arthritis
4. other conditions (such as osteomyelitis, tuberculosis, and tumor) that affect their walking function; had a contraindication to exercise; and exhibited cognitive impairment

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | one month
  Pain intensity will be measured by visual analogue scale (VAS).
static balance | one month
  static balance will be measured by Postural stability test by Biodex balance SD.
Dynamic balance | one month
  Dynamic balance will be measured by Limit of stability Test by biodex balance SD.
.Functional abilities | one month
  Functional abilities will be measured by Arabic- language version of knee injury and osteoarthritis outcome score physical function short form (KOOS-PS).

CONTACTS AND LOCATIONS:
Locations (1):
- Mti University, Cairo, Egypt